CLINICAL TRIAL: NCT06683456
Title: EMOTE: a Smartphone Application for Binge Eating Based on DBT Skills: a Randomized Controlled Trial
Brief Title: EMOTE: a Smartphone Application for Binge Eating Based on DBT Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPCEUP/RH5
Record Dates: First submitted 2024-07-29; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Binge Eating
Keywords: DBT; Binge Eating; Feeding and Eating Disorders; Application
MeSH Terms: conditions — Bulimia; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eMOTE (Experimental): Participants will have access to eMOTE for eight weeks.
  Interventions: Behavioral: eMOTE
- Waiting List (No Intervention): Participants will be on a waiting list group for eight weeks. After that period, the participants will have access to eMOTE.

INTERVENTIONS:
Behavioral: eMOTE — The intervention combines psychoeducation, mindfulness skills, emotion regulation skills, and distress tolerance skills, along with self-monitoring of meals, behaviours and feelings.
  Arms: eMOTE

SUMMARY:
Binge eating, whether formally diagnosed or occurring at subthreshold levels, is associated with adverse health consequences and decreased quality of life.

Access to accessible, cost-effective interventions that effectively address binge eating episodes is critical for individuals with this condition, and smartphone applications have demonstrated promise in treating binge eating and related disorders.

This study aims to evaluate the efficacy of eMOTE, a novel smartphone application for binge eating based on Dialectical Behavior Therapy (DBT) skills. For this purpose, a randomized controlled trial will be conducted in which women who self-report binge eating episodes will be randomly assigned to the app intervention group or a waiting list group.

DETAILED DESCRIPTION:
eMOTE is a self-help application for women struggling with binge eating episodes. The application was developed based on DBT skills and has four modules: psychoeducation, mindfulness skills, emotion regulation skills, and distress tolerance skills. Additionally, it includes two self-monitoring diaries that allow the input of data related to food, behaviors, feelings, and exercises. The application content will be delivered through text, audios, and videos.

For this study, adult individuals with binge eating episodes who are fluent in Portuguese and own a smartphone will be recruited. The recruitment will be conducted through social media, the University of Porto, and other relevant institutions.

Participants who enrol in eMOTE will be required to fill out online self-report instruments and provide their body mass index (BMI) at baseline (T0), two months (T1), and four months after randomization (T2). A researcher not involved in the study will conduct the randomization process.

Participants will be randomly allocated to two groups: the experimental and control groups. In the experimental group, the participants will have access to eMOTE for eight weeks, while in the control group, the participants will be on a waiting list for eight weeks, and after this period, the participants will have access to eMOTE. The investigators will analyze the changes in the frequency of objective and subjective binge eating episodes, eating disorder psychopathology, BMI, intuitive eating, depression, anxiety, stress, compensatory behaviors, mindfulness, and difficulties in emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* female;
* aged 18 years or older;
* self-report at least one binge eating episode over the past four weeks;
* owned a smartphone;
* fluent in Portuguese.

Exclusion Criteria:

* attending psychotherapy (face-to-face or digital) or another clinical trial;
* body mass index below 18.5;
* self-report an average of eight or more episodes of binge eating or inappropriate compensatory behaviours per week;
* being pregnant;
* self-report bipolar disorder, psychotic disorder, substance abuse, suicidal ideation or borderline personality disorder.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes in binge eating symptoms | From Baseline to 2-months follow-up
  Assessed by Binge Eating Scale - BES. The Binge Eating Scale (BES) is a 16-item self-report questionnaire used to assess the presence and severity of binge eating behaviors. The scale's total score can range from 0 to 46, with higher scores indicating more severe levels of binge eating.
Changes in objective binge eating episodes | From Baseline to 2-months follow-up
  Assessed by Eating Disorder Examination Questionnaire - EDE-Q. The Eating Disorder Examination Questionnaire (EDE-Q) is a 36-item self-report tool designed to assess the range, frequency, and severity of behaviors associated with eating disorder diagnoses. The total score on the EDE-Q can range from 0 to 6, with higher scores indicating more severe eating difficulties.

SECONDARY OUTCOMES:
Changes in BMI | From Baseline to 2-months follow-up
  Assessed by a Body Composition Analyzer
Changes in intuitive eating | From Baseline to 2-months follow-up
  Assessed by Intuitive Eating Scale-2 - IES-2. The Intuitive Eating Scale-2 (IES-2) includes 23 items assessing various dimensions of intuitive eating. The total score on the IES-2 can range from 1 to 5, with higher scores indicate a greater tendency toward intuitive eating behaviors.
Changes in depression, anxiety and stress | From Baseline to 2-months follow-up
  Assessed by Depression, Anxiety and Stress Scale - 21 - DASS-21. The Depression Anxiety Stress Scales-21 (DASS-21) is a 21-item self-report questionnaire designed to measure levels of depression, anxiety, and stress. The scale provides three scores, one for each subscale, where the minimum is 0 and the maximum is 21, with higher scores indicate greater severity of emotional distress in each of these areas.
Changes in eating disorder psychopathology | From Baseline to 2-months follow-up
  Assessed by Eating Disorder Examination Questionnaire - EDE-Q. The Eating Disorder Examination Questionnaire (EDE-Q) is a 36-item self-report tool designed to assess the range, frequency, and severity of behaviors associated with eating disorder diagnoses. The total score on the EDE-Q can range from 0 to 6, with higher scores indicating more severe eating difficulties.
Changes in subjective binge eating episodes | From Baseline to 2-months follow-up
  Assessed by Eating Disorder Examination Questionnaire - EDE-Q. The Eating Disorder Examination Questionnaire (EDE-Q) is a 36-item self-report tool designed to assess the range, frequency, and severity of behaviors associated with eating disorder diagnoses. The total score on the EDE-Q can range from 0 to 6, with higher scores indicating more severe eating difficulties.
Changes in compensatory behaviors | From Baseline to 2-months follow-up
  Assessed by Eating Disorder Examination Questionnaire - EDE-Q. The Eating Disorder Examination Questionnaire (EDE-Q) is a 36-item self-report tool designed to assess the range, frequency, and severity of behaviors associated with eating disorder diagnoses. The total score on the EDE-Q can range from 0 to 6, with higher scores indicating more severe eating difficulties.
Acceptability | T1 - immediately after intervention
  Assessed by utility and satisfaction with the digital intervention. Participants will rate the usefulness of each module and their satisfaction with it, using a scale from 1 to 5, ranging from "not at all" to "extremely".

OTHER OUTCOMES:
Changes in emotion regulation | From Baseline to 2-months follow-up
  Assessed by Difficulties in Emotion Regulation Scale - DERS. The Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report questionnaire designed to assess difficulties in emotional regulation. The total score on DERS can range from 36 to 180, with higher scores indicating greater difficulties in regulating emotions.
Changes in mindfulness | From Baseline to 2-months follow-up
  Assessed by Mindful Attention and Awareness Scale - MAAS. The Mindful Attention and Awareness Scale (MAAS) is a 15-item self-report instrument that measures the extent to which individuals act with awareness in daily life. The total score can range from 1 to 6, and higher scores indicate more mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Telma Cruz, MSc, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Psychology and Educational and Education Sciences, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No